CLINICAL TRIAL: NCT06065384
Title: Central and Peripheral Neuroplasticity in Cervical Spinal Cord Injury Following Intensive Upper Limb Motor Training
Brief Title: Neural Plasticity and Motor Recovery After Upper Extremity Motor Training in People With c-SCI
Acronym: REPAIR-SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Annemie Spooren (Other)
Collaborators: Research Foundation Flanders (Other); University of Aarhus (Other); University of Sydney (Other); University Hospital, Ghent (Other); Universitaire Ziekenhuizen KU Leuven (Other); Adelante, Centre of Expertise in Rehabilitation and Audiology (Other); Rehabilitation Hospital RevArte (Unknown)
Responsible Party: Sponsor-Investigator, Annemie Spooren, Prof. Annemie Spooren, Hasselt University
Organization: Hasselt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REPAIR-SCI_UH
Record Dates: First submitted 2023-06-14; First posted 2023-10-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord rehabilitation; therapy dose; neural plasticity; motor recovery; upper limb training
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensive upper limb training (Experimental): The intervention group receives 6 hours of motor training each week upon usual care during 8 weeks. This involves active and targeted motor training of all affected muscles below the injury level in the context of functional activities.
  Interventions: Other: experimental group: intensive motor training
- usual care (Other): The control group receives only standard rehabilitation and care
  Interventions: Other: usual care

INTERVENTIONS:
Other: experimental group: intensive motor training — Intervention group: receive an extra 6 hours of motor training each week (distributed over the week) for 8 weeks. It will involve active and targeted motor training of all affected muscles of the upper limb below the level of the injury within the context of practice of functional activities. Interventions will be goal directed and individualized to the needs of each participant with a focus on training that addresses each person's specific motor problem, promoting motor learning as well as stimulating neural plasticity. All patients will continue to receive usual physiotherapy and usual rehabilitation.
  Arms: intensive upper limb training
Other: usual care — usual rehabilitation
  Arms: usual care

SUMMARY:
After spinal cord injury (SCI), there is a disruption in neural circuits resulting in paralysis. There is not yet a cure for paralysis. In persons with Cervical SCI (pwC-SCI) recovery of arm-hand function is very important as it has a significant impact on the patients' level of independence and quality of life. Recovery is assumed to involve alterations in both central and peripheral motor systems. Motor training at an intensive dosage potentially provides a powerful stimulus for neurological recovery. This project exploits the peripheral and central neuroplastic effect of an early (<13 weeks after injury) and intensive (8 weeks of 6 hours in addition to usual care) upper limb motor training program (EIUMT) directed at recovery below the level of the injury in pwC-SCI within an international multi-center randomized controlled trial including 44 pwC-SCI. It has 4 objectives: to investigate 1)central neural plasticity by identifying alterations in cortical neuroplasticity and corticospinal excitability; 2)peripheral neural plasticity by identifying alterations in axonal excitability and number of motor units; 3)behavioral motor recovery of upper limb and 4)relationships between dose dimensions of motor intervention and behavioral and neurophysiological outcome measures after EIUMT. Cutting-edge neurophysiological measures are used to provide insight in the mechanism of neuroplasticity after EIUMT and will be taken before and after EIUMT and at 6 months follow-up.

DETAILED DESCRIPTION:
Background of the study:

Paralysis or paralysis is the most common effect of spinal cord injury (SCI) on individuals. Paralysis affects the ability to walk, perform self-care, live independently and participate in work and leisure activities. In individuals with cervical spinal cord injury, arm and hand function is very important. The most promising and easily implemented intervention that could promote neurological recovery and make a lasting difference in the lives of people with spinal cord injuries is early and intensive motor training aimed at recovery below the injury level. This intervention takes advantage of the early plasticity of the nervous system. By maximizing muscle activation in the first few weeks after injury, we can target the nervous system's unique capacity for neural plasticity where changes can occur in central and peripheral motor systems.

Objective of the study:

This project aims to investigate peripheral and central neuroplasticity following an early (<13 weeks after injury) and intensive (8 weeks of 6 hours of additional therapy) upper extremity motor training program (EIUMT) aimed at recovery below the lesion level. This project has 4 objectives: to investigate 1) central neural plasticity (identify changes in cortical neuroplasticity and corticospinal excitability; 2) peripheral neural plasticity (identify change in axonal excitability and number of motor units); 3) clinical motor recovery of the upper limbs and 4) relationships between dose dimensions of motor intervention and clinical and neurophysiological outcome measures after EIUMT. Advanced neurophysiological measurements and clinical measurements will be taken before and after EIUMT and at 6-month follow-up.

Study design:

a multicenter pragmatic randomised controlled study in 2 countries

Study population:

44 persons with cervical spinal cord injury (22 participants in the control and intervention groups) Inclusion criteria: Individuals are eligible to participate if they have suffered a traumatic or non-traumatic cervical spinal cord injury within the previous 13 weeks, have AIS (ASIA Impairment Scale) A lesion with motor function more than three levels below motor level (on one or both sides) or have AIS C or AIS D lesion (as defined by the International Standards for the Neurological Classification of spinal cord injury), are older than 16 years of age, have received permission to begin rehabilitation and are likely to remain an inpatient for the next 8 weeks.

Exclusion criteria: Participants will be excluded if they have a significant medical or physical condition or psychiatric illness that could prevent the person from participating in the study or would place the person at unacceptable risk if they were to participate.

Intervention:

The intervention group receives 6 hours of motor training each week. This involves active and targeted motor training of all affected muscles below the injury level in the context of functional activities.

The control group receives only standard rehabilitation and care.

Primary study parameters/outcome of the study (Baseline vs 8 weeks after randomisation):

Central plasticity via: Single pulse TMS (transcranial magnetic stimulation) (Resting Motor Threshold) Peripheral plasticity via: Peripheral nerve assessment (Compound muscle action potential (CMAP)) Functional recovery via: Grades redefined assessment of strength, sensibility and Prehension (GRASSP)

Secondary study parameters/outcome of the study:

Clinical Measures: Upper Extremity Motor Score, Spinal Cord Independence Measure (SClM-selfcare); Van Lieshout Test (VLT); Hand-Held Dynamometry; accelerometry (session density: active therapy time/session length); perceived difficulty and exertion) Central plasticity: Single Pulse TMS: Stimulus-Response Function, Cortical mapping, Paired pulse TMS: SICI (short interval intracortical inhibition); LICI (long interval intracortical inhibition) Peripheral plasticity: NET (Nerve excitability testing) and MScanFit MUNE.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non-traumatic C-SCI in the preceding 13 weeks; age over 16 years; have an incomplete SCI categorized as AIS C or D or an AIS A SCI with zones of partial motor paralysis (as defined by the International Standards for the Neurological Classification of SCI (ISNCI) and medically stable.

Exclusion Criteria:

* SCI with ASIA Impairment Scale (AIS) A without zones of partial preservation (decided based on former studies) and expertise of the team; SCI with any significant medical condition that could prevent the person from participating. Patients will be excluded from the measures of central plasticity in the presence of contraindications for TMS application such as epilepsy, metal implants in the brain, defibrillator, pacemaker, and pregnancy

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-08-28 (Estimated)

PRIMARY OUTCOMES:
changes in single pulse TMS: resting motor threshold | - before intervention; at 4 weeks (inbetween measure), at 8 weeks (after intervention) and at 6 months follow-up
  to asses changes in cortical reactivity
Changes in Compound Muscle Action Potential (CMAP) | - before intervention; at 4 weeks (inbetween measure), at 8 weeks (after intervention) and at 6 months follow-up
  Changes in amplitude of CMAP
changes in GRASSP | - before intervention; at 8 weeks (after intervention) and at 6 months follow-up
  Grades redefined assessment of strength sensibility and Prehension

SECONDARY OUTCOMES:
Single-pulse TMS: Stimulus Response Curve | - before intervention; at 4 weeks (inbetween measure), at 8 weeks (after intervention) and at 6 months follow-up
  - to assess cortical excitability
changes SICI | - before intervention; at 8 weeks (after intervention) and at 6 months follow-up
  to evaluatie changes in Short interval intracortical inhibition
changes in LICI | - before intervention; at 8 weeks (after intervention) and at 6 months follow-up
  long-interval intracortical inhibition
changes in MscanFit MUNE | - before intervention; at 4 weeks (inbetween measure), at 8 weeks (after intervention) and at 6 months follow-up
  Compound muscle action potential (CMAP) scans will be recorded
changes in single pulse TMS: mapping | - before intervention; at 8 weeks (after intervention) and at 6 months follow-up
  to evaluate changes in cortical reorganisation
changes in NET (Nerve excitability testing) | - before intervention; at 4 weeks (inbetween measure), at 8 weeks (after intervention) and at 6 months follow-up
  Stimulus-Response Curve, Strength duration time constant (SDTC), threshold electrotonus (TE), I/V relationship (I/V) and recovery cycles (RC) will be measured.
changes in behavioral measures: Upper extremity motor score | - before intervention; at 8 weeks (after intervention) and at 6 months follow-up
  score on 50
changes in Spinal Cord independence Measures | - before intervention; at 8 weeks (after intervention) and at 6 months follow-up
  questionaire: self-care score
changes in Van Lieshout Test | - before intervention; at 8 weeks (after intervention) and at 6 months follow-up
  basis upper extremity skills
changes in hand held dynamometry | - before intervention; at 8 weeks (after intervention) and at 6 months follow-up
  strength in hand
Goal satisfaction | - before intervention; at 8 weeks (after intervention) and at 6 months follow-up
  Subjective scoring 0-10 of four goals

OTHER OUTCOMES:
Subjectively perceived session difficulty | measurement of one week during the 2., 5. and 8. week of intervention duration; before and after completion of session
  VAS
Objective active time | - measurement of one week during the 2., 5. and 8. week of intervention duration
  accelerometry
Subjectively perceived session intensity | measurement of one week during the 2., 5. and 8. week of intervention duration; before and after completion of session
  VAS (perceived exertion)
Therapy documentation | whole trial period of 8 weeks
  Total session length and UL training session length based on therapy documentation

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Spooren, Prof. Dr., Principal Investigator — Hasselt University
Locations (4):
- Belgium (3):
  - Revalidatieziekenhuis RevArte, Antwerp
  - UZGent, Ghent
  - UZLeuven Campus Pellenberg, Leuven
- Zorggroep Adelante, Hoensbroek, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Pseudomised data will be discussed with Aarhus University because they will assist in data analyses.
  The protocol will be shared with the partners (Aarhus University, Sydney University, UZ Gent, UZ Leuven, RZ RevArte, and Adelante Zorggroep)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: during and after data gathering
Access Criteria: only for collaborating partners